CLINICAL TRIAL: NCT00934882
Title: Phase I, Open-label, Non-placebo Controlled Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of BAY73-4506 in Combination With mFOLFOX6 or FOLFIRI as First or Second Line Therapy in Patients With Metastatic Colorectal.
Brief Title: Study to Determine Safety, Pharmacokinetics, Pharmacodynamics of BAY73-4506 in Combination With mFOLFOX6 or FOLFIRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11656; 2008-007151-27 (EudraCT Number)
Record Dates: First submitted 2009-07-03; First posted 2009-07-08 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer; Targeted therapy; Multi-kinase inhibitor; FOLFOX; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — Administration of the multi-kinase inhibitor BAY73-4506 (160 mg once daily from Day 4 to Day 10 and from Day 18 to Day 24) as oral treatment in combination with the chemotherapy regimen mFOLFOX6 or FOLFIRI in patients with metastatic Colorectal Cancer

SUMMARY:
This multi-center, open-label, non-randomized, non-placebo-controlled, Phase I study will define the safety profile and tumor response profile of the multi-kinase inhibitor BAY73-4506 as oral treatment in combination with the chemotherapy regimen mFOLFOX6 or FOLFIRI in patients with metastatic CRC. It will also determine the impact of the combined administration on the concentration of drugs over time (pharmacokinetics) of BAY73-4506, oxaliplatin, 5 FU, and irinotecan.

This study will be conducted at approximately 5 - 8 study centers in Germany. Up to 60 patients will be enrolled into this study to ensute that at least 12 - 15 patients for each combination regimen can be evaluated for safety and pharmacokinetics. For this reason a minimum of 20 patients will receive mFOLFOX6 in combination with BAY73-4506 and at least 20 patients will receive FOLFIRI in combination with BAY73-4506.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum.
* At least 1 measurable lesion as per RECIST
* ECOG Performance Status of 0 - 1
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* More than 1 previous chemotherapy for Colorectal Cancer. Adjuvant chemotherapy for Colorectal Cancer (Stage I, II, II) is permitted, if the adjuvant therapy ended >6 month before screening.
* Previous FOLFOX treatment for patients who will be included in the mFOLFOX6 cohort apart from FOLFOX treatment in an adjuvant setting.
* Previous FOLFIRI treatment for patients who will be included in the FOLFIRI cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event Collection | 3 years
Effect of BAY73-4506 on the pharmacokinetics of mFOLFOX6 and FOLFIRI (Cmax, AUC, through concentration of BAY73-4506 and Cmax, AUC of Platinum, Irinotecan and its metabolite SN-38, 5-Flourouracil) | Cycle 1 and Cycle 2

SECONDARY OUTCOMES:
Biomarker status | Screening, Cycle 1, Cycle 2, Cycle 3
Pharmacodynamic parameters | 3 years
Tumor response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Germany (7):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Oldenburg, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia
  - Dresden, Saxony

REFERENCES:
- [Result] Schultheis B, Folprecht G, Kuhlmann J, Ehrenberg R, Hacker UT, Kohne CH, Kornacker M, Boix O, Lettieri J, Krauss J, Fischer R, Hamann S, Strumberg D, Mross KB. Regorafenib in combination with FOLFOX or FOLFIRI as first- or second-line treatment of colorectal cancer: results of a multicenter, phase Ib study. Ann Oncol. 2013 Jun;24(6):1560-7. doi: 10.1093/annonc/mdt056. Epub 2013 Mar 13. PMID 23493136